CLINICAL TRIAL: NCT06507150
Title: AI-assisted Migraine Education: Efficacy, Safety and Patients' Acceptance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Chiara Zecca, Prof, dr, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EOC.NSI.HA.2401
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIME - AI-assisted migraine education (Experimental): Intervention group: it receives AI-assisted migraine education in addition to standard migraine education
  Interventions: Other: AI-assisted migraine education (AIME)
- SME -Standard Migraine Education (No Intervention): Control group: it receives standard migraine education only

INTERVENTIONS:
Other: AI-assisted migraine education (AIME) — AIME Group will undergo the established migraine education plus AI-assisted education.
  Arms: AIME - AI-assisted migraine education

SUMMARY:
Migraine affects 1 in 7 people globally, significantly impacting quality of life and economic productivity. Despite its prevalence, limited awareness leads to misdiagnosis, inadequate treatment, and stigmatization. AI can enhance migraine management through improved diagnosis, prediction, and personalized education. The primary objective of this study is to determine if adding AI-assisted migraine education to standard education improves patients' understanding of their condition more effectively.

DETAILED DESCRIPTION:
Migraine affecting approximately 1 in 7 individuals globally, significantly impacts quality of life and economic productivity due to its associated healthcare and social burdens. Despite its prevalence, awareness and understanding of migraine remain limited, contributing to misdiagnosis, inadequate treatment, and the perpetuation of stigmatization.

Artificial Intelligence (AI) may advance migraine management by improving diagnosis, prediction, and educational outreach. AI applications are currently being employed in diagnosing migraines more accurately by analyzing comprehensive patient data, thus differentiating migraine from other types of headaches. Additionally, AI algorithms predict migraine episodes, enabling preemptive measures. They also streamline medication management through reminders and monitor patient adherence, which is crucial for preventing medication overuse and optimizing treatment outcomes.

Moreover, AI can bridge the educational gap in migraine understanding. By using adaptive learning technologies, AI platforms can deliver personalized educational content, tailored to an individual's knowledge level and learning pace, enhancing understanding and engagement. This approach not only facilitates better management of the condition but also promotes a broader societal awareness essential for destigmatizing migraine.

The primary objective of this study is to ascertain if the addition of AI-assisted migraine education to standard migraine education yields a superior improvement in the patients' understanding of their condition.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years at the time of signing the informed consent
* Newly diagnosis of migraine, confirmed through the medical chart
* The participant must be capable of giving signed informed consent
* Access to a laptop, computer, smartphone, or tablet

Exclusion Criteria:

* Insufficient knowledge of the protocol language (italian)
* Patients with cognitive impairment and/or unable to use or access the AI-powered learning platform developed in this study.
* Vulnerable participants (e.g. minors, participants incapable of judgment or participants under tutelage)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to ascertain if the addition of AI-assisted migraine education to standard migraine education yields a superior improvement in the patients' understanding of their condition. | 3 months
  Difference in the proportion of correct responses to a set of 20 migraine-related questions via the Migraine Intel Quotient test score (MiQ score) between Standard Migraine Education (SME Group) and the AI-assisted migraine education added to Standard Migraine Education (AIME group) at 3 months after baseline.

SECONDARY OUTCOMES:
Investigate if the two types of educations have persistent effect over time up to 6 months. | 6 months
  To assess changes in the MiQ score from baseline to 3 months and to 6 months, and from 3 months to 6 months in the SME group and AIME group.
Evaluate the participants' subjective perception of each education experience | 6 months
  To report patients' evaluation of learning experience at 3 and 6 months after baseline in both SME and AIME groups by 10 Visual Analog Scale (VAS) scoring, and comparison between groups at each timepoint
Investigate migraine clinical course following either education interventions | 6 months
  To assess changes in the number of monthly migraine days, migraine intensity, and migraine duration as well as the HIT-6 and MIDAS scores at 3 and 6 months after baseline in SME and AIME groups, and between SME and AIME groups at each time point.
Evaluate the frequency and the quality of adverse events (AEs) occurring during education interventions | 6 months
  To describe frequency and type of AEs occurring during the study period in SME and AIME groups.education interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Ente Ospedaliero Cantonale - Ospedale Regionale di Lugano, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided